CLINICAL TRIAL: NCT06932939
Title: Comparison of Two Caries Risk Assessment Tools CAMBRA123 Versus (CAT) AAPD Among a Group of Egyptian Children: A Cross- Sectional Study
Brief Title: Comparison of CAMBRA123 and AAPD (CAT) for Caries Risk in Egyptian Children
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hanaa AlKarib, principal investigator, Cairo University
Other Study IDs: CTCRATCVA-AAGOEC-2025
Record Dates: First submitted 2025-04-10; First posted 2025-04-17 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Caries Experience

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study goal is to compare two indices in Egyptian children aged 3-6 years in caries detection and time needed for assessment which will contribute to variable data for pediatric oral health assessment locally and globally.

DETAILED DESCRIPTION:
This study will ensure that patients receive precise evaluations and guide early, appropriate preventive measures or treatments. Over time, this will contribute to reducing caries progression and related complications. Also, Parents become more aware of their children's dental health status, emphasizing the importance of early detection and intervention. Furthermore, Comparing the indices will provide insights into which tool is most efficient and reliable for detecting caries in children 3-6 years old.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3 to 6 years.
* Both genders.
* No underlying medical conditions affecting oral health.

Exclusion Criteria:

* Uncooperative patient.
* Children with cognitive impairments that prevent understanding the study procedures.
* Parents refused.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: This study will be conducted at the outpatient clinics of the Pediatric and Dental Public Health Department among group of (3-6) years old- Faculty of Dentistry, Cairo University - Egypt.
Sampling Method: Non-Probability Sample
Enrollment: 376 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Caries risk assessment using AAPD | baseline (single visit)
  Caries risk will be categorized as Low, Moderate, or High based on the American Academy of Pediatric Dentistry (AAPD) criteria.
  * Unit of Measure: Category (Low / Moderate / High)
Caries risk assessment using CAMBRA123 | baseline (single visit)
  Caries risk will be evaluated using the CAMBRA 123 scoring system, which assigns scores from -4 to +18, categorized as:
  * Low: -4 to -1
  * Moderate: 0 to +3
  * High: +4 to +13
  * Very High: +14 to +18

SECONDARY OUTCOMES:
Time For index Application | baseline (single visit)
  The time required to apply each caries assessment index (CAMBRA123 and AAPD) will be measured in seconds for each child during the clinical examination

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry Cairo University, Cairo, Giza Governorate, Egypt

REFERENCES:
- [Background] Featherstone JDB, Crystal YO, Alston P, Chaffee BW, Domejean S, Rechmann P, Zhan L, Ramos-Gomez F. A Comparison of Four Caries Risk Assessment Methods. Front Oral Health. 2021 Apr 28;2:656558. doi: 10.3389/froh.2021.656558. eCollection 2021. PMID 35048004
- [Background] Devraj IM, Shankaraguru GM, Jairam LS, Dhull KS, Bhojraj N. Comparison of two different caries risk assessment tools for infants and toddlers - A cross-sectional study. J Indian Soc Pedod Prev Dent. 2024 Jan 1;42(1):9-14. doi: 10.4103/jisppd.jisppd_546_23. Epub 2024 Apr 15. PMID 38616421